CLINICAL TRIAL: NCT03844009
Title: Impact of Computer Debriefing During Screen-based Simulation of Neonatal Resuscitation
Brief Title: Computer Debriefing and Screen-based Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilumens (Other)
Responsible Party: Principal Investigator, Daphne Michelet, Principal Investigator, Ilumens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RNN
Record Dates: First submitted 2019-02-07; First posted 2019-02-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Computer Simulation; Neonatal Resuscitation

STUDY DESIGN:
Intervention Model Description: randomized controlled study comparing two groups, one intervention group (debriefing) and one control group (no debriefing)
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor (questionnaire) was blinded of the allocation group of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debriefing (Experimental): Participant's of the debriefing group had a computer integrated debriefing at the end of each scenario of the computer-based simulator
  Interventions: Other: Computer integrated debriefing
- No debriefing (No Intervention): Participant's of the debriefing group had no computer integrated debriefing at the end of each scenario of the computer-based simulator

INTERVENTIONS:
Other: Computer integrated debriefing — At the end of each computer-based simulation, the participant had a computer integrated debriefing of his performance during the neonatal resuscitation simulation and a debriefing based on an auto-evaluation of his non-technical skills.
  Arms: Debriefing

SUMMARY:
Debriefing after simulation plays a crucial role in student learning and medical practice. This paper focuses on impact of computer debriefing technique on knowledge retention of midwives during screen-based simulation of neonatal resuscitation.

DETAILED DESCRIPTION:
Simulation, including screen-based simulation, is employed in medicine to enhance competency and improve care. It has been practiced for centuries in its primitive form as uses of wax Venus or obstetrics dolls to teaching anatomical knowledge or know-how/gestures. Many benefits come from simulations as the capacity to practiced procedures without any risk to the patient, the possibility of trainees to commit errors and learn from these errors, the repeatability of scenario that can be different or presented to learners many times, and then the opportunity to improved technical and non-technical skills among learners. Specifically, screen-based simulation has many advantages as portability (easy to move), distribution and replicability (usable by many learners at differences places in the world), repeatability (people not faced frequently in their regular practice), even be remotely usable. Screen-based simulation appears in literature to be a complement of mannequin simulation. Indeed, since last years the development of computer science has made it possible to create new kind of simulators in the medical field for the acquisition of knowledge, know-how and technical gestures, more realistic and interactively rich.

Debriefing is considered as a part of simulation-based training and cannot be separated of simulators. Debriefing improve professional practice, clinical skills and competences. It exists different debriefing methods: post simulation debriefing, in-simulation debriefing, verbal instructor debriefing, video-assisted instructor debriefing, self-debriefing or also multimedia debriefing. However, debriefing is considered by many as a communication between student/learner and teacher, after a situation (e.g. simulation), and about this experience. It is not just a feedback on performance but also a communication process about the impact of the experience or performance explanation.

This study aims to evaluate the impact of a computer integrated debriefing of technical and non-technical skills on retention and performance of neonatal resuscitation management by trainee's midwives.

Thirty student in midwifery in fourth year will participate. The study protocol is the following:

Baseline knowledge questionnaire, randomization of the participants. Day one: Tutorial of the simulator, First scenario (+/- debriefing depending of the allocation group), second scenario (+/- debriefing depending of the allocation group).

Day two (two month later): knowledge questionnaire, tutorial of the simulator, one scenario (+/- debriefing depending of the allocation group).

ELIGIBILITY:
Inclusion Criteria:

* Student in midwifery in fourth year in france (penultimate year of the midwifery studies)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
knowledge retention | two months
  Knowledge assesment based on a validated questionnaire created from International Liaison Committee On Resuscitation guidelines at T0 (before simulation), T1 (after the first simulation session) and T2 (after the second simulation session, two month later)

SECONDARY OUTCOMES:
Non-technical skills assesment | two months
  Evaluation of the Anesthetist Non technical skills score at T1 (first session) and T2 (second session, two month later)
Technical skills assessment | two months
  Evaluation of the Modified Neonatal Resuscitation Program Evaluation score at T1 (first session) and T2 (second session, two month later)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Tesnière, PhD, Study Director — Ilumens
Locations (1):
- Ilumens, Paris Descartes University, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Heide PA, van Toledo-Eppinga L, van der Heide M, van der Lee JH. Assessment of neonatal resuscitation skills: a reliable and valid scoring system. Resuscitation. 2006 Nov;71(2):212-21. doi: 10.1016/j.resuscitation.2006.04.009. Epub 2006 Sep 20. PMID 16987590
- [Background] Donoghue A, Nishisaki A, Sutton R, Hales R, Boulet J. Reliability and validity of a scoring instrument for clinical performance during Pediatric Advanced Life Support simulation scenarios. Resuscitation. 2010 Mar;81(3):331-6. doi: 10.1016/j.resuscitation.2009.11.011. Epub 2010 Jan 4. PMID 20047787
- [Derived] Michelet D, Barre J, Truchot J, Piot MA, Cabon P, Tesniere A. Effect of Computer Debriefing on Acquisition and Retention of Learning After Screen-Based Simulation of Neonatal Resuscitation: Randomized Controlled Trial. JMIR Serious Games. 2020 Aug 11;8(3):e18633. doi: 10.2196/18633. PMID 32780021